CLINICAL TRIAL: NCT03809702
Title: Efficacy of Pregabalin for the Treatment of Acute Herpetic Neuralgia and for the Prevention of Post Herpetic Neuralgia- a Randomized Controlled Trial
Brief Title: Efficacy of Pregabalin for the Treatment of Acute Herpetic Neuralgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Collaborators: University Grants Commission (Other)
Responsible Party: Principal Investigator, Dr Suchana Marahatta, Associate Professor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPKoirala
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; Herpetic neuralgia; Pregabalin
MeSH Terms: conditions — Herpes Zoster | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin group (Active Comparator): Group 1: Pregabalin tablet 75 mg orally twice daily for 4 weeks will be given to the subjects in this group along with other routine treatment Here, the intervention is administration of Pregabalin tablet 75 mg
  Interventions: Drug: Pregabalin
- Placebo group (Placebo Comparator): Group 2: Placebo tablet twice daily for 4 weeks will be given to the subjects in this group along with other routine treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pain score in group 1 (intervention group) will be compared with pain score in group 2 (placebo group)
  Arms: Pregabalin group
Drug: Placebo — Pain score in group 1 (intervention group) will be compared with pain score in group 2 (placebo group)
  Arms: Placebo group

SUMMARY:
All eligible Herpes Zoster patients will be randomized into two groups. Group 1 will be the treatment group receiving Pregabalin 75 mg twice daily for 4 weeks in addition to other routine treatment. Whereas, group 2 will be the control group receiving all routine treatment similar to group 1 except Pregabalin. Instead control group will receive Placebo.

DETAILED DESCRIPTION:
This study wants to see the role of Pregabalin in acute herpetic neuralgia pain reduction and for the prevention of post herpetic neuralgia incidence as compared to placebo group. For this purpose, all eligible Herpes Zoster patients will be randomized into two groups (41 patients in each group i.e.82 total patients). Group 1 will be the treatment group receiving Pregabalin 75 mg twice daily for 4 weeks in addition to other routine treatment. Whereas, group 2 will be the control group receiving all routine treatment similar to group 1 except Pregabalin. Instead of pregabalin, control group will receive Placebo. The pain will be evaluated in all patients in each follow visits (weekly follow up for 4 weeks then monthly follow up for next three months). If it is difficult for the patient to present physically, telephonic follow up will be done to find the pain score in the required time. Also, DLQI (Dermatological life quality index) will be assessed at the first and last visit of the patient.

At the end, pain score will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of HZ presenting within 72 hours of onset of rash,
* With pain score 40 or above on 100 mm pain Visual Analogue Scale at the screening visit,
* Giving written consent for the study.
* Age between 18-70 years

Exclusion Criteria:

* HZ presenting after 72 hours of onset
* Pain score less than 40 at baseline
* Who took the stable doses of oral analgesics like: NSAIDs, acetaminophen, opioids and antidepressant within six hours of screening visit
* Using Pregabalin and Gabapentin within last 72 hours
* Nerve block therapy within the last 48 hours
* History of hypersensitivity to the drug or its ingredients
* Use of topical medications within 12 hours
* Unable to come for follow up because of severe systemic illness
* Significant hepatic and renal disease,
* Bed ridden patients or those who are physically unfit for follow up visits.
* Ethically considered vulnerable members- pregnant/lactating mothers/newborn/children below 12 years /physically or mentally challenged individuals/HIV/ AIDS/IV drug users

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage reduction of visual analogue scale (VAS) of pain in each visit in intervention and placebo group | Eight months
  Percentage reduction of visual analogue scale (VAS) of pain in each follow up visits in intervention group as compared to the placebo group

SECONDARY OUTCOMES:
Prevention of Post Herpetic Neuralgia | 12 months
  Incidence of post herpetic neuralgia in pregabalin group and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Suchana Marahatta, MBBS, MD, Principal Investigator — B.P. Koirala Institute of Health Sciences
Locations (1):
- B P Koirala Institute of Health Sciences, Dharān, Koshi, Nepal